CLINICAL TRIAL: NCT02674308
Title: Entyvio (Vedolizumab) Long-term Safety Study: An International Observational Prospective Cohort Study Comparing Vedolizumab to Other Biologic Agents in Patients With Ulcerative Colitis or Crohn's Disease
Brief Title: Entyvio (Vedolizumab) Long Term Safety Study
Acronym: Entyvio PASS
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: MLN-0002_401; MLN0002-401 (Other: Secondary Sponsor Identification Number)
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Ulcerative Colitis and Crohn's Disease
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vedolizumab
  Interventions: Drug: Vedolizumab
- Other Biologic Agents
  Interventions: Other: Other Biologic Agents

INTERVENTIONS:
Drug: Vedolizumab
  Groups: Vedolizumab
Other: Other Biologic Agents — Other biologic agents include: Adalimumab, Certolizumab pegol, Golimumab, and Infliximab
  Groups: Other Biologic Agents

SUMMARY:
The purpose of this study is to assess the long-term safety of vedolizumab versus other biologic agents in participants with Ulcerative Colitis (UC) or Crohn's Disease (CD).

DETAILED DESCRIPTION:
The drug being tested in this prospective, observational study is called vedolizumab. Vedolizumab is being used to treat people who have UC or CD. This study will look at the long-term safety of vedolizumab versus other biologic agents in participants with UC or CD. The study will enroll approximately 5000 participants. All participants enrolled in this will belong to one of the two treatment group:

* Vedolizumab
* Other Biologic Agents -adalimumab, certolizumab pegol.

Golimumab and infliximab. Study drugs will be prescribed by the physician according to local prescribing information in the participating countries. This multi-centre trial will be conducted worldwide. The overall time to participate in this study is 7 years. Participants will make visits at every 6 months to their treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, by the participant or a legally acceptable representative.
2. Aged at least 18 years.
3. Initiating vedolizumab or another biologic agent for UC or CD.
4. Signed release form, by the participant or a legally acceptable representative, permitting abstraction of the participant's medical records at Baseline and during participation in the study.

Exclusion Criteria:

1. The participant is enrolled in a clinical trial in which treatment for CD or UC is managed through a protocol.
2. Prior treatment with vedolizumab.
3. Any other reason that, in the Investigator's opinion, makes the participant unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with ulcerative colitis (UC) or Crohn's disease (CD) who are initiating Entyvio or another biologic agent. Participants may be biologic-naive or have prior use of a biologic agent
Sampling Method: Probability Sample
Enrollment: 5302 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events of Special Interest | 7 years
  Adverse events of special interest in this study includes serious and opportunistic infections, gastrointestinal infections, respiratory infections, other clinically significant infections: malignancies; infusion-related reactions and hypersensitivity, hepatic injury; psoriasis and other skin events, other SAEs and adverse reactions.

SECONDARY OUTCOMES:
Disease Severity in Ulcerative Colitis (UC) Participants | Baseline and at every 6 months (up to 7 years)
  Disease severity will be measured using the Mayo score for ulcerative colitis and is ranged from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores: stool frequency, rectal bleeding and physician rating of disease activity, each ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe).
Disease Severity in Crohn's Disease (CD) Participants | Baseline and at every 6 months (up to 7 years)
  Disease severity will be measured using the Harvey-Bradshaw Index (HBI) for crohn's disease. HBI is used in the assessment and quantification of symptoms and the present level of disease activity of participants with Crohn's disease. It is a validated clinical index for Crohn's disease,HBI score consists of clinical parameters of general well-being (0= very well 1=slightly below average, 2=poor, 3=very poor, 4=terrible); abdominal pain (0=none, 1=mild, 2=moderate, 3=severe); number of liquid stools per day; abdominal mass (0=none, 1=dubious, 2=definite, 3=tender); and complications (8 items: arthralgia, uveitis, erythema nodosum, aphthous ulcers, pyoderma gangrenosum, anal fissures, new fistula, abscess [score 1 per item]).Lower scores indicate better well-being. The scores are classified as: <5=remission, 5-7=mild disease, 8-16=moderate disease and >16=severe disease. Minimum score is 0 and no pre-specified maximum score as it depends on the number of liquid stools.
Participant Reported Quality of Life Assessment Using Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | Baseline and at every 6 months (up to 7 years)
  The Short IBD Questionnaire is an instrument used to assess quality of life and is a disease-specific health-related quality of life questionnaire, that consists of 10 questions, each question is scored on a scale from 1 (poor quality of life) to 7 (good quality of life). The scores are summed up and divided by 10 for a mean score ranging from 1 (poor quality of life) to 7 (good quality of life). A higher score indicates a better health-related quality of life.
Participant Reported Quality of Life Assessment Using 12-Item Short Form Health Survey (SF-12) | Baseline and at every 6 months (up to 7 years)
  The SF-12 health questionnaire is a 12 question assessment of functional health and well-being. The survey asks about various health aspects, including physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health (psychological distress and psychological well-being). Two summary measures are derived: the Physical and the Mental Health Component Summary. For each component summary, survey items were weighted and summed to create a summary score between 0 and 100 with higher score indicating better quality of life.
Time to Treatment Discontinuation | Baseline and at every 6 months (up to 7 years)
  Time to discontinuation for Entyvio and the other biologic agents will be measured.
Reasons for Treatment Discontinuation | Baseline and at every 6 months (up to 7 years)
  Reasons for discontinuations for Entyvio and the other biologic agents will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (287):
- United States (66):
  - University of Alabama, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - University of Arizona Medical Center, Tucson, Arizona
  - Scripps Clinic, La Jolla, California
  - Stanford University, Palo Alto, California
  - South Bay Gastroenterology Medical Group, Torrance, California
  - Gastroenterology Center of Connecticut P.C., Hamden, Connecticut
  - Middlesex Gastroenterology Associates, Llc, Middletown, Connecticut
  - Gastroenterology Group of Naples, Naples, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Gulf Region Clinical Research Institute, Pensacola, Florida
  - Emory University Hospital, the Emory Clinic, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Atlanta Gastroenterology Associates, Suwanee, Georgia
  - Illinois Gastroenterology Groupllc Northwest Gastroenterologists, Arlington Heights, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Northshore University Health Systems, Evanston, Illinois
  - Loyola University, Maywood, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - Kansas Gastroenterology, Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - New Orleans Research Institute, Metairie, Louisiana
  - Louisiana Research Center, Llc, Shreveport, Louisiana
  - Crohn'S and Colitis Center, Boston, Massachusetts
  - Boston University Moakley Building Center For Digestive Disorders, Boston, Massachusetts
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Infusion Associates, Grand Rapids, Grand Rapids, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Digestive Health Center, Pa, Ocean Spring, Mississippi
  - St. Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Chi Health Alegent Creighton Clinic, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Englewood Endoscopic Associates, Englewood, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saratoga-Schenectady Gastroenterology Associates, Burnt Hills, New York
  - Digestive Disease Center, Fishkill, New York
  - Northwell Health, Great Neck, New York
  - Nyu Langone Long Island Clinical Research Associates, Great Neck, New York
  - Nyu Langone Medical Center, New York, New York
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Gastroenterology Group of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Trihealth Digestive Institute, Cincinnati, Ohio
  - Mark Osterman, Philadelphia, Pennsylvania
  - Philadelphia Va Medical Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Consultants in Gastroenterology - Columbia, Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Fort Sam Houston, Texas
  - Baylor University Medical Center, Houston, Texas
  - Ut Health Science Center, Houston, Texas
  - Spring Gastroenterology, Humble, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Austria (8):
  - Krankenhaus Der Elisabethinen Linz Gmbh, Oberosterreich
  - Kh Der Barmherzigen Schwestern, Ried im Innkreis
  - Ordination Dr. Thomas Haas Darmpraxis Salzburg, Salzburg
  - Salk Salzburg, Salzburg
  - Landesklinikum St. Poelten, Sankt Pölten
  - Medizinischen Universitat Wien - Allgemeines Krankenhaus (Akh) - Universitaetsklinik Fuer Innere Medizin Iii, Vienna
  - Loha For Life, Vienna
  - KH WELS, Wels
- Belgium (23):
  - Olv Aalst - Gastro-Enterologie, Aalst
  - Imelda - Gastro-Enterologie, Bonheiden
  - Chu Saint Pierre - Service de Gastroenterologie, Brussels
  - Cub Hopital Erasme, Brussels
  - HIS-IZZ, Brussels
  - Uz Brussel - Gastro-Enterologie, Brussels
  - Uz Antwerpen - Gastro-Enterologie, Edegem
  - Ziekenhuis Oost Limburg - Gastro-Enterologie, Genk
  - Az Maria Middelares - Gastro-Enterologie, Ghent
  - Az St Lucas - Gastro-Enterologie, Ghent
  - Uz Gent - Gastro-Enterologie, Ghent
  - Jessa Ziekenhus - Gastro-Enterologie, Hasselt
  - Az Groeninge - Campus Kennedylaan - Gastro-Enterologie, Kortrijk
  - Universitaire Ziekenhuizen (Uz) Leuven - Gasthuisberg, Leuven
  - Centre Hospitalier Chretien (Chc) - Clinique Saint-Joseph (Hopital St-Joseph) - Gastro-Enterologie, Liège
  - Chr de La Citadelle, Liège
  - Chu Liege - Gastro-Enterologie, Liège
  - Az Sint Maarten, Campus Rooienberg, Mechelen
  - Chu Ambroise-Pare, Mons
  - Clinique Et Maternite Sainte-Elisabeth, Namur
  - Clinique St Pierre Asbl, Ottignies
  - Az Delta - Gastro-Enterologie, Roeselare
  - Centre Hospitalier de Wallonie Picardie, Site Notre Dame, Tournai
- Canada (7):
  - Okanagan Clinical Trials Ltd., Kelowna, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - McMasters University, Hamilton, Ontario
  - Scott Shulman Medical Prof. Corp, North Bay, Ontario
  - Taunton Surgical Centre-Oshawa Clinic, Oshawa, Ontario
  - University of Toronto - St. Michaels Hospital, Toronto, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
- Croatia (4):
  - University Hospital Center Osijek, Osijek
  - Clinical Hospital Centre Split, Split
  - Kbc Split, Split
  - University Hospital Dubrava, Zagreb
- Denmark (6):
  - University Hospital, Aalborg, Aalborg
  - Rigshospitalet, Abdominal Centre, Copenhagen
  - Bispebjerg Univarsity Hospital, Copenhagen NV
  - Hvidovre Hospital, Hvidovre
  - Nykobing Falster Sygehus, Nykøbing Falster
  - Silkeborg Hospital, Silkeborg
- Estonia (3):
  - West-Tallinn Central Hospital (Ltkh), Tallinn
  - North Estonian Regional Hospital, Tallinn
  - Tartu University Hospital, Tartu
- France (24):
  - Chu Amiens Picardie - Service Hepato-Gastro-Enterologie, Amiens
  - C H U Angers, Angers
  - Hopital Avicenne, Bobigny
  - Centre Hospitalier Universitaire (Chu) de Caen - Service D'Hepatogastroenterologie, Caen
  - C.H.U de Tours - Hopital Trousseau, Chambray-lès-Tours
  - Chu de Clermont Ferrand - Hopital Estaing, Clermont-Ferrand
  - Hopitaux Civils de Colmar, Colmar
  - Centre Hospitalier Regional Universitaire (Chru) de Lille - Hopital Claude Huriez, Lille
  - Hospices Civils de Lyon (Hcl) - Hopital Edouard Herriot, Lyon
  - Chu Hopital Nord, Marseille - Service D'Hepato-Gastro-Enterologie, Marseille
  - University Hospital St Eloi, Montpellier
  - Centre Hospitalier Universitaire (Chu) de Nice - Hopital L'Archet 2 - Pole Digestif, Nice
  - Chu Nimes - Hopital Caremeau, Nîmes
  - Centre Hospitalo Universitaire (Chu) - Hopital Saint-Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hopital Du Haut Leveque - Service D'Hepato-Gastro-Enterologie Et Nutritution, Unite de Soin Normalise, Pessac
  - Hospices Civils de Lyon (Hcl) - Centre Hospitalier Lyon-Sud - Hepatogastroenterologie, Pierre-Bénite
  - Centre Hospitalier Annecy Genevois, Pringy
  - Chu de Reims - Hopital Robert Debre, Reims
  - Centre Hospitalier Universitaire (Chu) de Rouen, Rouen
  - Service Gastro-Enterologie Hopital Nord - Chu de Saint Etienne, Saint-Etienne
  - Hopital Rangueil - Service de Gastroenterologie, Toulouse
  - Ch Gustave Dron - Hopital de Tourcoing, Tourcoing
  - Ch Valenciennes - Hopital Jean Bernard - Service Maladies de L'Appareil Digestif Et de La Nutrition, Valenciennes
- Germany (46):
  - Praxis Dr. Med. Eberhard Meier, Amberg
  - Charite Campus Campus Mitte, Berlin
  - Praxis Dr. Mross, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin (Cbf) - Medizinische Klinik I, Berlin
  - Charite Campus Virchow Klinikum - Medizinische Klinik Mit Schwerpunkt Hepatologie Und Gastroenterologie, Berlin
  - Praxis Fur Gastroenterologie Am Bayerischen Platz, Berlin
  - Sana Klinik Biberach, Biberach
  - Medizinisches Versorgungszentrum (Mvz) Dachau, Dachau
  - Stadtisches Klinikum Dessau, DESSAU-ROsLAU
  - Technische Universitaet Dresden - Universitaetklinikum Carl Gustav Carus - Medizinische Klinik Und Poliklinik I, Dresden
  - Universitatsklinikum Erlangen Medizinische Klinik I - Studien Ambulanz Ced, Erlangen
  - St. Josef Krankenhaus Essen-Werden / Abteilung Fur Gastroenterologie, Essen
  - Agaplesion Markus Krankenhaus, Medizinische Klinik 1, Frankfurt
  - Crohn-Colitis Centrum Rhein-Main, Frankfurt am Main
  - Praxis Dr. Med. Thomas Zeisler, Halle
  - Krankenhaus Martha-Maria Halle Dolau Ggmbii, Klinik Fur Innere Medizin I, Halle
  - Universitatsklinik Und Poliklinik Fur Innere Medizin I, Halle
  - Asklepios Westklinikum Hamburg, Hamburg
  - Hafced E.K., Hamburg Eppendorf
  - Universitatsklinikum Heidelberg, Heidelberg
  - Praxis Fur Gastroenterologie, Heidelberg
  - Gastroenterologische Gemeinschaftspraxis Dr. Felten, Herne
  - Praxis Group, Jerichow
  - PRAXIS, Köthen
  - Eugastro Gmbh, Leipzig
  - Universitat Leipzig, Medizinische Fakultat, Leipzig
  - Gesellschaft Fuer Klinische Studien, Leipzig
  - St. Marien Krankenhauses - Medizinischen Klinik I, Ludwigshafen am Rhein
  - Staedtisches Klinikum Luneburg, Lüneburg
  - Universitatsklinikum Magdeburg A. O. R. - Klinik Fur Gastroenterologie, Magdeburg
  - Universitaetsmedizin Mainz, I.Med.Klinik, Geb.605, Eg, Zi.0240, Mainz
  - Gastroenterologische Schwerpunkt Praxis, Mannheim
  - Praxis Dr. Krammer, Mannheim
  - Universitaetsklinikum Mannheim (Umm) - Ii Medizinische Klinik, Mannheim
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Klinikum Der Universitat Munchen, München
  - Medizinische Versorgungszentrum Portal 10, Münster
  - Gastroenterologische Fachpraxis Am Germania Campus, Münster
  - Praxis Group, Nuremberg
  - Praxiszentrum Alte Malzerei, Regensburg
  - Eric Norgaard Jorgensen, Remscheid
  - Gpr Mvz Gastroenterologie, Rüsselsheim am Main
  - Gemeinschaftspraxis - Endoskopiezentrum M. Hasenstein, Saarbrücken
  - Gastroenterologische Gemeinschaftspraxis - Stade, Stade
  - Uni-Klinik Tubingen, Tübingen
  - Gastro Data Gbr, Wiesbaden
- Greece (7):
  - University and General Hospital of Alexandroupoli, Alexandroupoli
  - General Hospital of Athens 'Evangelismos', Athens
  - General and University Hospital of Western Athens 'Attiko', Athens
  - St. Panteleimon General Hospital of Nikaia, Athens
  - University and General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina - Division of Gastroenterology, Ioannina
  - Theagenio Hospital of Thessaloniki, Thessaloniki
- Ireland (6):
  - Mercy University Hospital Cork, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St James Hospital, Dublin
  - St. Vincent'S University Hospital, Dublin
  - National University of Ireland Galway, Galway
- Israel (11):
  - Haemek Medical Center, Afula
  - Soroka University Medical Center (Sumc), Beersheba
  - Rambam Health Care Campus (Rhcc) - Institute of Gastroenterology, Haifa
  - Bnai Zion Mc, Haifa
  - Clalit Health Services - Lev Talpiot, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Tel Aviv University - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Clalit Medical Services - Migdal Hamea, Tel Aviv
  - Maccabi Healthcare Services, Tel Aviv
  - Tel Aviv Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center (Ahmc) - Institute of Gastroenterology, Zrifin
- Italy (24):
  - Ospedale Civile Giuseppe Moscati, Avellino Campania
  - Spedali Civili Gastroenterology Unit University of Brescia, Brescia
  - Fondazione Poliambulanza, Brescia
  - Azienda Ospedaliera Per Lemergenza Cannizzaro, Catania
  - Azienda Ospedaliero-Universitaria Careggi (Aouc), Florence
  - Casa Sollievo Della Sofferenza, Foggia
  - Ospedale Morgagni Pierantoni Forli U.O. Gastroenterologia Ed Endoscopia, Forlì
  - Policlinico G Martino, Messina
  - A.O. Guido Salvini Di Garbagnate Milanese, Milan
  - Fondazione Irccs Ca' Granda Osp Magg Policlinico, Milan
  - Asst Fatebenefratelli Sacco, Milan
  - Universita Federico Ii, Napoli
  - Ospedale Maggiore Della Carita, Novara
  - Policlicnico Universita Paolo Giaccone, Palermo
  - Ao San Camillo Forlanini, Roma
  - Ospedale Nuovo Regina Margherita, Roma
  - Ospedale Sandro Pertini, Roma
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Ospedale San Filippo Neri, Roma
  - Universita Campus Bio-Medico, Rome
  - Policlinico Tor Vergata, Rome
  - Universita Di Salerno Aou San Giovanni Di Dio E Ruggi D'Aragona, Salerno
  - Ao Ordine Mauriziano Di Torino, Torino
  - Osp Di Circolo Fondazione Macchi, Varese
- Netherlands (7):
  - VUMC, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum - Mdl, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Erasmus Mc, Rotterdam
  - Zuyderland, Sittard
- Norway (4):
  - Nordlandssykehuset Hf Bodo, Bodø
  - Sykehuset Innlandet Hf Hamar, Hamar
  - Akershus University Hospital, Nordbyhagen
  - Oslo Univeristy Hospital Ulleval Hospital, Oslo
- Instituto Portugues de Oncologia de Lisboa Francisco Gentil, Epe, Lisbon, Portugal
- Slovenia (2):
  - General Hospital Celje, Celje
  - University Medical Center Maribor, Maribor
- Spain (6):
  - Hospital Univ. Germans Trias I Pujol, Badalona
  - Hospital de Bellvitge, Hospitalet
  - Hospital Universitario La Paz, Madrid
  - Complexo H. Pontevedra-Hospital de Montecelo, Pontevedra
  - Consorci Sanitari de Terrassa, Terrassa
  - H. Alvaro Cunqueiro, Vigo
- Sweden (3):
  - Medical Dept, Gastroenterology Unit, Stockholm
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Danderyds Sjukhus Ab, Stockholm
- Switzerland (4):
  - Universitaetsspital Bern - Inselspital - Universitaetsklinik Fuer Viszerale Chirurgie Und Medizin (Uvcm) - Klinik Und Poliklinik Fuer Gastroenterologie, Bern
  - Gastroenterologische Praxis Balsiger, Seibold & Partner Crohn-Colitis-Zentrum Hochhaus Lindenhofspital, Bern
  - Kantonsspital St. Gallen - Gastroenterologie, Sankt Gallen
  - Universitatspital Zurich, Zurich
- United Kingdom (25):
  - Nevill Hall Hospital - Aneurin Bevan Health Board, Abergavenny
  - Blackpool Victoria Hospital (Bvh) - Gastroenterology Department, Blackpool
  - Bradford Teaching Hospitals, Bradford
  - Frimley Park Hospital, Camberley
  - University Hospitals Coventry and Warwickshire Nhs Trust - University Hospital (Walsgrave Hospital), Coventry
  - Derby Hospitals Nhs Foundation Trust - Royal Derby Hospital (Derby City General Hospital), Derby
  - The North West London Hospitals Nhs Trust (Nwlh) - St Mark'S Hospital, Harrow
  - Hull and East Yorkshire Nhs Trust, Hull
  - Airedale Nhs Foundation Trust, Keighley
  - Forth Valley Royal Hospital, Larbert
  - Royal Liverpool University Hospital, Liverpool
  - Barts Health Nhs Trust, London
  - Nhs Foundation Trust - Homerton University Hospital (Huh), London
  - King'S College Hospital (Kch) Nhs Foundation Trust, London
  - Manchester Royal Infirmary, Manchester
  - Royal Gwent Hospital, Newport
  - The University of Nottingham - Nottingham Digestive Diseases Centre (Nddc) (Wolfson Digestive Diseases Centre), Nottingham
  - Salford Royal Nhs Foundation Trust, Salford
  - University of Sheffield - Sheffield Teaching Hospitals Nhs Foundation Trust - Royal Hallamshire Hospital (Rhh), Sheffield
  - The Shrewsbury and Telford Hospital Nhs Trust - Royal Shrewsbury Hospital, Shrewsbury
  - University Hospital Southampton Nhs Foundation Trust, Southampton
  - Pinderfields Hospital - Mid Yorkshire Hospital Trust, Wakefield
  - Nhs Trust - Weston Area Health - Weston General Hospital, Weston-super-Mare
  - The Royal Wolverhampton Hospitals Nhs Trust - New Cross Hospital, Wolverhampton
  - Western Sussex Hospitals Nhs Trust - Worthing Hospital, Worthing

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60274db2bf003ab498b5?idFilter=%5B%22MLN-0002_401%22%5D